CLINICAL TRIAL: NCT01348113
Title: Efficacy of a Brief Alcohol Intervention for Non Dependant Alcohol-misusing Patients Undergoing a Scheduled Surgery: a Randomized Controlled Trial
Brief Title: Efficacy of a Brief Alcohol Intervention for Non Dependant Alcohol-misusing Patients Undergoing a Scheduled Surgery
Acronym: ITBCHIR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RCB 2009-A00591-56; PHRC/09-09 (Other: Rennes University Hospital)
Record Dates: First submitted 2010-07-02; First posted 2011-05-05 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Alcohol Abuse; Alcohol Problem; AOD Misuse
Keywords: Alcohol Use Disorders Identification Test; alcohol dependence; Alcohol problem
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders | interventions — Ethanol; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Alcohol Intervention (Experimental)
  Interventions: Other: Brief Alcohol intervention
- No intervention (No Intervention)

INTERVENTIONS:
Other: Brief Alcohol intervention — Brief intervention consists typically in a brief assessment, giving patients personal feedback, dealing with resistance and ambivalence, establishing a goal of reduced alcohol use, and giving a workbook; reinforcement visits or calls are included.
  Other Names: BAI
  Arms: Brief Alcohol Intervention

SUMMARY:
Excessive alcohol consumption is a worldwide major public health problem. Brief interventions have shown to be an efficient treatment modality for problem drinkers, but have never been tested in scheduled surgery.

Patients will be recruited in various surgery units in 7 hospital in France. All patients attending a scheduled surgery will be screened during the visit with the anaesthesist by the Alcohol Use Disorders Identification Test (AUDIT). Patients aged 30-75 with an AUDIT between 7 and 12, corresponding to at risk or harmful use, will be proposed to enter a control study and randomized between a brief intervention by a trained nurse during the post-surgery hospitalisation and no intervention. Twelve months after the surgery, a research technician will interview by telephone patients and evaluate AUDIT and alcohol consumption of the last month.

DETAILED DESCRIPTION:
Excessive alcohol consumption is a worldwide major public health problem. Persons who drink more than 2-3 drinks per day are at risk for numerous medical, psychological and social problems. Brief interventions have shown to be an efficient treatment modality for problem drinkers in settings such as primary care, emergencies or psychiatric hospitals by numerous randomized studies. Brief intervention consists typically in a brief assessment, giving patients personal feedback, dealing with resistance and ambivalence, establishing a goal of reduced alcohol use, and giving a workbook; reinforcement visits or calls are included. Brief interventions seem to be particularly effective in patients with alcohol problem without dependence.

Screening for alcohol problem is best done using standardized questionnaires, as the Alcohol Use Disorders Identification Test (AUDIT), developed by WHO and translated in many languages. The AUDIT allows distinguishing between normal alcohol use, harmful or at risk use and dependence and is easy to use.

No study on brief intervention has been conducted in scheduled surgery. This seems to be a promising situation, since there is first a visit with the anaesthetist, during which screening for alcohol problem should occur, then a hospitalisation, during which the intervention could be made. It is possible that patients are more concerned by their health when they come to hospital for a surgery.

The aim of this controlled, randomized study is to test the hypothesis that a brief intervention, consisting in a visit with a trained nurse, followed by a telephone call three months later, in patients with at risk or harmful alcohol use, undergoing a scheduled surgery, could be efficient to promote the decrease of alcohol consumption.

Patients will be screened during the visit with the anaesthetist with AUDIT. Patients with AUDIT between 7 and 12 will be proposed to enter the study, and randomised between Brief Intervention and no intervention. A research technician will interview patients 12 months after the surgery, with assessment of the AUDIT and alcohol consumption. CDT and GGT will be measured prior to surgery, then at 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Aged 30 to 75 years old
* With a scheduled surgery
* Presenting an Alcohol Use Disorders Identification Test score between 7 and 12 (included) during the routine visit with the anaesthesist prior to hospitalisation
* Being capable of understanding the information note
* Who gave a written informed consent
* Affiliated to a medical insurance

Non inclusion Criteria:

* Surgery in relation to alcohol consumption (chronic pancreatitis, oropharyngeal cancer for example) or modifying alcohol consumption (liver transplantation for example),
* No telephone number
* Dependence to alcohol (Alcohol Use Disorders Identification Test score ≥ 13)
* History of alcohol weaning complications
* History of addiction care
* Life expectancy less than 5 years
* Decompensated psychiatric disease
* Usual consumption (more than three times a week) of illicit products
* Person deprived of freedom or under guardianship
* Participation or intent to participate in another biomedical research

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Rate of patients getting back to an Alcohol Use Disorders Identification Test score <7 | 1 year

SECONDARY OUTCOMES:
Evolution of the Alcohol Use Disorders Identification Test score | 1 year
Alcohol consumption in the month preceding the final evaluation at 1 year | 1 year
Gamma-GT and CDT evolution | 1 year
Frequency of normalization of gamma-GT and CDT measures | 1 year
Rate of patients in the Brief Alcohol Intervention group getting back to an Alcohol Use Disorders Identification Test score <7, with stratification on the Prochaska score | 1 year
Feeling of the patients towards the Brief Alcohol Intervention | 1 year
  recollection, acceptability, relevance, recollection of the recall at 3 months, acceptability of the recall at 3 months
Prevalence of alcohol misuse, with or without dependence, in patients seen in pre-anaesthesia consultation | 6 months
Proportion of total population presenting an increase in gamma-GT and CDT in comparison with upper limits of normal | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Romain MOIRAND, MD, PhD, Principal Investigator — Rennes University Hospital; Jean-Michel REYMANN, PhD, Study Chair — Rennes University Hospital
Locations (1):
- Unité d'Alcoologie et Hépatologie Générale, Département d'Anesthésie Réanimation- Hôpital de Pontchaillou, Rennes, France